CLINICAL TRIAL: NCT06826833
Title: Efficacy of Erector Spinae Plane Block in Flexible Ureterorenoscopy (URS) Surgery: A Randomized Controlled Trial
Brief Title: ESP Block for Postoperative Analgesia in URS Surgery
Acronym: ESPURS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Onur Baran, Asst. Prof., Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNKU-URS001
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Analgesia; Postoperative Pain Management; Nephrolithiasis
MeSH Terms: conditions — Agnosia; Nephrolithiasis | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESP Block Group (Experimental): A regional anesthesia technique in which 20 mL of 0.25% bupivacaine is injected under ultrasound guidance at the T8-T10 level to provide postoperative pain relief.
  Interventions: Procedure: Erector Spinae Plane (ESP) Block
- Control Group (No Intervention): Patients will receive routine multimodal analgesia without an ESP block.

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) Block — A regional anesthesia technique in which 20 mL of 0.25% bupivacaine is injected under ultrasound guidance at the T8-T10 level to provide postoperative pain relief.
  Arms: ESP Block Group

SUMMARY:
The goal of this clinical trial is to determine whether the erector spinae plane (ESP) block provides better pain relief after flexible ureterorenoscopy (URS) surgery compared to standard analgesia alone. Researchers want to know:

Does the ESP block reduce pain levels in the first 24 hours after surgery?

Does it lower the need for opioid pain medication?

Does it reduce the need for additional (rescue) pain treatment?

Does it decrease the likelihood of postoperative nausea and vomiting (PONV)?

Participants will be randomly placed into one of two groups:

ESP Block Group: Participants will receive an ESP block using 20 mL of 0.25% bupivacaine under ultrasound guidance before surgery.

Control Group: Participants will receive standard pain management without a nerve block.

All participants will receive general anesthesia during surgery and multimodal pain management after surgery. Researchers will compare pain scores, opioid use, rescue analgesic needs, and the occurrence of nausea and vomiting between the two groups.

DETAILED DESCRIPTION:
Intervention Group (ESP Block): Patients will receive 20 mL of 0.25% bupivacaine (1:1 diluted with 0.5% bupivacaine) under ultrasound guidance at the T8-T10 level.

Control Group: No block will be performed, and patients will receive standard postoperative multimodal analgesia.

Procedure Description: The ESP block will be performed under sterile conditions with a high-frequency linear ultrasound probe. A 100-mm echogenic needle will be inserted in a cephalocaudal direction to deposit the local anesthetic deep to the erector spinae muscle at the transverse process level. The correct spread of the anesthetic will be confirmed via real-time ultrasound imaging.

All patients will receive standardized general anesthesia and multimodal analgesia.

Outcome measures include postoperative pain (NRS), opioid consumption, rescue analgesia requirement, and postoperative nausea and vomiting (PONV).

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective flexible ureterorenoscopy (URS).

Age: 18-65 years.

ASA I-II.

Willing to participate and provide written informed consent.

Exclusion Criteria:

BMI >35 kg/m².

Allergy to local anesthetics.

Coagulation disorders or use of anticoagulants.

Patients requiring emergency surgery.

Patients with infection at the ESP block site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Numeric Rating Scale - NRS) | 0, 2, 6, 12, 24 hours postoperatively.
  The Numeric Rating Scale (NRS, 0-10) will be used to assess postoperative pain intensity. Participants will be asked to rate their pain on a scale from 0 to 10, where:
  * 0 = No pain
  * 10 = Worst possible pain

SECONDARY OUTCOMES:
Total Opioid Consumption (IV PCA Morphine Equivalent) | From 0 hours (postoperatively) to 24 hours postoperatively, assessed at 0, 2, 6, 12, and 24 hours.
  Description: Total opioid consumption will be recorded in morphine milligram equivalents (MME) administered via IV patient-controlled analgesia (PCA).
Postoperative Nausea and Vomiting (PONV) | From 0 hours (postoperatively) to 24 hours postoperatively, assessed at 0, 2, 6, 12, and 24 hours.
  The incidence of postoperative nausea and vomiting (PONV) will be recorded, defined as nausea and/or vomiting requiring treatment with ondansetron IV.
Pain-Free Duration | From the end of surgery until the first request for pain medication, assessed up to 24 hours postoperatively.
  Pain-free duration is defined as the time from the end of surgery to the first request for analgesia (when the patient reports pain requiring medication).

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Şahin, Assoc. Prof., Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdağ Namık Kemal University Research Hospital, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Bryniarski P, Bialka S, Kepinski M, Szelka-Urbanczyk A, Paradysz A, Misiolek H. Erector Spinae Plane Block for Perioperative Analgesia after Percutaneous Nephrolithotomy. Int J Environ Res Public Health. 2021 Mar 31;18(7):3625. doi: 10.3390/ijerph18073625. PMID 33807296
- See also: Ref. 2 — https://doi.org/10.1097/AAP.0000000000000451